CLINICAL TRIAL: NCT02584556
Title: A Randomized Controlled Trial of Radical Hepatectomy With Adjuvant Transcatheter Arterial Chemoembolization Versus Adjuvant Systemic Chemotherapy for Hepatocellular Carcinoma
Brief Title: Adjuvant Transcatheter Arterial Chemoembolization Versus Adjuvant Systemic Chemotherapy for Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Chengcheng Liao, Director, Principal Investigator, Clinical Professor, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TA-C/hcc
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- systemic chemotherapy (Experimental): Pirarubicin(Brand Name:Pirarubicin - Main Luck Pharmaceutical, China) 30mg/m2 intravenously on Day 1 and Oxaliplatin(Brand Name: Eloxatin) 100 mg/m2 intravenously on Day 2 every 3 weeks within 4-6 weeks after hepatic resection(a total of 4 cycles).
  Interventions: Drug: systemic chemotherapy
- Transcatheter Arterial Chemoembolization (Active Comparator): Transcatheter Arterial Chemoembolization (Lipiodol 5-10ml,Pirarubicin17mg/m2 and Oxaliplatin 30mg/m2 are infused through the right and left hepatic arteries,followed by embolization using gelatin sponge particles(Gelfoam; Guangzhou)) within 4-6 weeks after hepatic resection(a total of 1 cycle).
  Interventions: Drug: Transcatheter Arterial Chemoembolization

INTERVENTIONS:
Drug: systemic chemotherapy — Pirarubicin(Brand Name:Pirarubicin - Main Luck Pharmaceutical, China) 30mg/m2 intravenously on Day 1 and Oxaliplatin(Brand Name: Eloxatin) 100 mg/m2 intravenously on Day 2 every 3 weeks starting 4-6 weeks after hepatic resection.
  Arms: systemic chemotherapy
Drug: Transcatheter Arterial Chemoembolization — Lipiodol 5-10ml,Pirarubicin17mg/m2 and Oxaliplatin 30mg/m2 are infused through the right and left hepatic arteries,followed by embolization using gelatin sponge particles(Gelfoam; Guangzhou) starting 4-6 weeks after hepatic resection.
  Arms: Transcatheter Arterial Chemoembolization

SUMMARY:
The purpose of this study is to determine that adjuvant systemic chemotherapy is superior to adjuvant transcatheter arterial chemoembolization(TACE) in prolonging recurrence free survival（RFS） in patients after radical resection of hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. a preoperative diagnosis of HCC with no previous treatment;
2. compensated cirrhosis with Child-Pugh class A, B or no cirrhosis;
3. multiple tumors more than 5 cm or tumor involving a major branch (the Wrstor second branch) of the portal or hepatic vein(s) on preoperative investigations, and on intraoperative ultrasonography and gross examination of the liver during operation;
4. on exploration and intraoperative ultrasonography, the tumor with multiple lesions localized in right or left hemiliver,or the main tumor localized in one lobe only with a small solitary lesion in contralateral lobe, or tumor involving a major branch (the Wrst or second branch) of the portal or hepatic vein(s), which could be safely resected without grossly remaining tumors, and the patient was judged to have well preserved liver function to survive the operation.
5. Adequate organ and marrow function, with neutrophil count≥1.5X10e9/L, platelet count≥75×10e9/L, AST or ALT﹤2.5×upper limit of normal (ULN), total bilirubin<1.5×ULN, international normalized ratio <1.5;normal baseline left ventricular ejection fraction_lower limit of normal for the institution. Patients with AST and ALT<5 ×ULN could be recruited if total bilirubin was in the normal range.

Exclusion Criteria:

1. documented allergy to study drugs; any previous TACE or systemic chemotherapy treatment before random assignment;
2. concomitant use of any other anticancer therapy, including interferon alfa and herbal medicine approved by the local authority to be used as anticancer medicine (except palliative radiotherapy to a nontarget lesion);
3. CNS metastasis;
4. Other serious illness or medical condition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
recurrence free survival | 6 months

SECONDARY OUTCOMES:
Overall survival | 3 months and 24 months
Time to Recurrence | 6 months and 12 months
Time to Recurrence within liver | 3 months and 12 months
Time of tumor distant metastasis | 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lequn Li, PhD, Study Director — Affiliated Tumor Hospital, Guangxi Medical University

REFERENCES:
- [Background] Zhong C, Guo RP, Li JQ, Shi M, Wei W, Chen MS, Zhang YQ. A randomized controlled trial of hepatectomy with adjuvant transcatheter arterial chemoembolization versus hepatectomy alone for Stage III A hepatocellular carcinoma. J Cancer Res Clin Oncol. 2009 Oct;135(10):1437-45. doi: 10.1007/s00432-009-0588-2. Epub 2009 May 1. PMID 19408012
- [Background] Peng BG, He Q, Li JP, Zhou F. Adjuvant transcatheter arterial chemoembolization improves efficacy of hepatectomy for patients with hepatocellular carcinoma and portal vein tumor thrombus. Am J Surg. 2009 Sep;198(3):313-8. doi: 10.1016/j.amjsurg.2008.09.026. Epub 2009 Mar 12. PMID 19285298
- [Background] Qin S, Bai Y, Lim HY, Thongprasert S, Chao Y, Fan J, Yang TS, Bhudhisawasdi V, Kang WK, Zhou Y, Lee JH, Sun Y. Randomized, multicenter, open-label study of oxaliplatin plus fluorouracil/leucovorin versus doxorubicin as palliative chemotherapy in patients with advanced hepatocellular carcinoma from Asia. J Clin Oncol. 2013 Oct 1;31(28):3501-8. doi: 10.1200/JCO.2012.44.5643. Epub 2013 Aug 26. PMID 23980077